CLINICAL TRIAL: NCT02176109
Title: Rôle Pronostique Des métabolismes du Stress Oxydatif et du Fer Dans Les Leucémies Aiguës Myéloblastiques
Brief Title: Metabolism Des LAM
Acronym: LAM-ROS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: gre-lam-fer; Métabolismes des LAM (Registry Identifier: 2013-A00762-43)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Iron; Acute Myeloid Leukemia; Diagnosis; Oxydative Stress
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — leukemic cells in order to rna and proteins study medullar plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, the investigators study the prognostic role of oxidative stress metabolism and iron in Acute myeloid leukemia.

DETAILED DESCRIPTION:
Primary goal of this study is to Evaluate the characteristics of regulatory networks of iron and redox balance in leukemic cells, to study the correlations between the prognosis of AML patients (in terms of response to induction chemotherapy and survival i) and metabolism of these markers. Secondary ones areto assess the impact of induction therapy on markers of oxidative stress and to correlate biological iron and redox metabolism with the molecular status of patients (eg Flt3/IDH/CEBPA/NPM...).

Eligibility criteria are patients at diagnostic of de novo acute myeloid leukemia (promyelocytic excluded) aged from 18 to 100 years.

ELIGIBILITY:
Inclusion Criteria:

de novo acute myeloid leukemic patient from 18 years to 99 years at diagnosis

Exclusion Criteria:

age under 18 years promelocytic leukemia secondary leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: de novo acute myeloid leukemic patient from 18 years to 99 years. promyelocytic leukemia excluded
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
overall survival Event-free survival Response to induction chemotherapy, overalll survival, event-free survival | five years after the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, Isere, France